CLINICAL TRIAL: NCT00690846
Title: A Multi-Center, Open Label Pilot Study to Determine the Safety and Efficacy of Adalimumab in the Treatment of Pyoderma Gangrenosum (HUM 04-37)
Brief Title: Study to Determine the Safety and Efficacy of Adalimumab in the Treatment of Pyoderma Gangrenosum
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Dr. Jorizzo has withdrawn from this study due to time it is taking to start
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002156; 32410
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2018-07

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): 40 mg weekly subcutaneous injection of adalimumab
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — 40 mg weekly adalimumab injection.
  Other Names: Humira

SUMMARY:
The purpose of this research study is to see if Humira (adalimumab) is effective and safe in the treatment of pyoderma gangrenosum.

DETAILED DESCRIPTION:
The primary objective of this study is to obtain preliminary data on the safety and efficacy of adalimumab for the treatment of PG. A secondary objective is to study gene expression in PG.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent.
* Subject is willing and able to participate in the study as an outpatient and is willing to comply with study requirements.
* Subject is 18 years of age or older.
* Subject has a diagnosis of pyoderma gangrenosum that involves total area of 3 cm2 or greater and is of sufficient severity to warrant systemic agents.
* If female of childbearing potential, subject will have a negative urine pregnancy test at Screening and Week 0.
* If female, subject will be either post-menopausal for > 1 year, surgically sterile (hysterectomy or bilateral tubal ligation), or practicing one form of birth control (abstinence, oral contraceptive, estrogen patch, implant contraception, injectable contraception, IUD, diaphragm, condom, sponge, spermicides, or vasectomy of partner). Female subjects will continue to use contraception for 6 months following the last injection.
* Screening laboratory results are within the following parameters:
* Subject has been on a stable dose of antibiotics, oral corticosteroids or other immunosuppressives, such cyclosporine, tacrolimus, azathioprine, methotrexate, or mycophenolate mofetil over the previous 4 weeks

Exclusion Criteria:

* Subject has evidence of a clinically significant, unstable or poorly controlled medical condition.
* Subject has a chest X-ray consistent with an active infection or previous exposure to TB and/or a positive purified protein derivative test at screening (>5 mm). (Subjects may participate if they are being actively treated in accordance with CDC guidelines.)
* Subject has a serious, active or recurrent bacterial, viral, or fungal infection. This includes hepatitis B and C, and HIV.
* Subject has been hospitalized for infection or received IV antibiotics within the previous 2 months prior to baseline.
* Subject has clinical evidence as determined by the investigator of acutely infected pyoderma gangrenosum or subject is receiving systemic antibiotics for the treatment of acute infection. Subjects receiving minocycline, tetracycline, dapsone, or other antibiotics for anti-inflammatory purposes are permitted.
* Subject has a history of tuberculosis without documented adequate therapy.
* Subject has a history of a central nervous system disorder/demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis.
* Subject has current signs or symptoms or history of systemic lupus erythematosus.
* Subject has been diagnosed with a malignancy within the past 5 years except for successfully treated non-melanoma skin cancer.
* Subject has signs or symptoms suggestive of a possible lymphoproliferative disease.
* Subject has a diagnosis of severe congestive heart failure (Class III or IV NYHA).
* Subject has had a substance abuse problem within the previous 3 years.
* Subject has been treated with an anti-TNF biologic immune response modifier, such as infliximab, adalimumab, or etanercept within the past 8 weeks.
* Subject has any dermatologic disease in the target site that may be exacerbated by treatment or interfere with examination.
* Subject has been administered an investigational drug in another clinical study within 30 days prior to baseline (or 5 half-lives, whichever is longer).
* Subject has a known allergy to adalimumab.
* Subject is female and is pregnant, is considering becoming pregnant during the study and for 6 months afterwards, or is nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07 (Estimated); Primary Completion 2007-07 (Estimated); Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
Mean change in the number of ulcers. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jorizzo, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States